CLINICAL TRIAL: NCT07196943
Title: Outcomes of Implant-Supported Equator Overdentures Following Fully Guided Static Implant Surgery: A Prospective Study
Brief Title: Prospective Outcomes of Guided Equator Overdentures
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Dr, Menoufia University
Other Study IDs: ADMNF-011225
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fully guided static computer-assisted implant surgery (CAIS) for mandibular overdentures using Equator® attachments — Mandibular edentulism will be rehabilitated with implant-supported overdentures using a fully guided static computer-assisted implant surgery (CAIS) protocol. Each patient will receive four implants placed in a quadrilateral configuration (lateral incisor and first premolar regions) under a stereolithographically manufactured surgical guide. Following 3-4 months of osseointegration, definitive mandibular overdentures will be fabricated and retained exclusively with Equator® attachment systems (Rhein 83, Bologna, Italy). Patients will be followed for 3 years to assess implant survival, peri-implant soft tissue health, and marginal bone changes.

SUMMARY:
This prospective clinical study evaluated the 3-year performance of mandibular implant-supported overdentures (IODs) placed using a fully guided static computer-assisted implant surgery (CAIS) protocol. Primary outcomes included implant survival, peri-implant soft tissue health, and marginal bone loss. Findings provide evidence for the predictability of digital surgical workflows in removable prosthodontics.

DETAILED DESCRIPTION:
Edentulism remains a prevalent global health concern that compromises oral function, esthetics, and quality of life. While conventional complete dentures are widely used, their limitations in mandibular stability often reduce patient satisfaction. Implant-supported overdentures (IODs) offer superior retention and function, but their long-term success depends heavily on precise implant placement.

Computer-assisted implant surgery (CAIS), particularly static fully guided protocols, has been shown to enhance surgical accuracy in fixed prosthodontics. However, evidence for their application in removable prosthodontics remains limited, despite the anatomical and prosthetic challenges often encountered in overdenture cases.

This prospective clinical study was designed to assess the 3-year clinical performance of mandibular IODs placed via a fully guided static CAIS workflow. Outcomes included implant survival, peri-implant soft tissue health, and marginal bone changes. The results provide valuable clinical insight into the role of digital surgical protocols in improving predictability and long-term success of overdenture rehabilitation.

ELIGIBILITY:
* Inclusion Criteria:

  * Completely edentulous mandible requiring implant-supported overdenture rehabilitation
  * Adequate bone volume to accommodate four implants in a quadrilateral configuration, confirmed by cone-beam computed tomography (CBCT)
  * Age between 40 and 75 years
  * Good general health with no systemic contraindications to implant surgery
  * Willingness and ability to provide informed consent
  * Commitment to attend all scheduled follow-up visits over the 3-year study period
* Exclusion Criteria:

  * Uncontrolled systemic diseases (e.g., diabetes mellitus, osteoporosis)
  * History of radiotherapy in the head and neck region
  * Untreated oral infections or severe periodontal disease
  * Poor oral hygiene or inability to comply with maintenance protocols
  * Heavy smoking (>10 cigarettes/day) or alcohol abuse
  * Known allergy or intolerance to materials or medications used in the study

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of completely edentulous adults aged 40-70 years, recruited from the outpatient clinic of [Institution Name]. All participants require mandibular implant-supported overdenture rehabilitation and have adequate bone volume to accommodate four implants in a quadrilateral configuration. Patients must be in good general health, able to provide informed consent, and committed to attending scheduled follow-up visits over the 3-year study period.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Implant Survival Rate | From prosthesis delivery to 36 months post-loading
  Defined as the percentage of implants remaining in function without mobility, pain, infection, or need for removal during the study period. Survival will be evaluated clinically at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El-Sawy, PhD, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Dentistry, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No
up on reasonable request from the corresponding author